CLINICAL TRIAL: NCT02488668
Title: Natural Sensory Feedback for Phantom Limb Modulation and Therapy
Brief Title: Surface Electrical Stimulation for Treatment of Phantom Limb Pain
Acronym: EPIONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winnie Jensen (Other)
Collaborators: Aalborg University Hospital (Other); University of Lausanne Hospitals (Other); University of Freiburg (Other); Université Montpellier (Other); Lund University (Other); Indiana University School of Medicine (Other); Novosense AB (Industry); Mxm-Obelia (Industry); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor-Investigator, Winnie Jensen, Professor, Aalborg University
Organization: Aalborg University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-602547-1; 602547 (Other Grant/Funding Number: FP7-HEALTH-2013-INNOVATION); NCT02519907 (obsolete NCT alias)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Phantom Limb Pain
Keywords: Transcutaneous Electrical Stimulation; Neuroplasticity; Sensory Feedback
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surface Electrical Stimulation (Experimental): Please see information under 'Detailed description'
  Interventions: Device: Surface Electrical Stimulation

INTERVENTIONS:
Device: Surface Electrical Stimulation — Surface electrical stimulation using the following devices; 1) INOMED surface stimulator, 2) The EPIONE Psychophysical Testing Platform software for stimulator control. Surface stimulation therapy is provided while providing visual guidance to the subject.

SUMMARY:
Phantom limb pain (PLP) is a frequent consequence of amputation, and it is notoriously difficult to treat. Amputation usually follows traumatic injuries or surgery following vascular diseases, diabetes, osteomyelitis or tumours in cases where the loss of the limb is required for the survival of the patient. The loss of a limb or other body parts is usually followed by the sensation that the lost body part is still present and can be felt. These phenomena are called, respectively, phantom awareness and phantom sensation. In 50-80% of amputees neuropathic pain develops in the lost limb also referred to as phantom limb pain (PLP). PLP can be related to a certain position or movement of the phantom limb, and might be elicited or worsened by a range of physical factors (e.g. changes in the weather or pressure on the residual limb) and psychological factors (e.g. emotional stress). It is well known that most treatments available for PLP today, such as pharmacological, surgical, anaesthetic, psychological and other, are ineffective.

Today it is believed that phantom limb pain may be related to changes in the cortex of the brain. There is evidence that these changes may be modulated - or even reversed - by providing sensory input to the stump or amputation zone. For example, cortical reorganization and alleviation of phantom limb pain has been observed in amputees following intense use of a hand prosthesis. However, there is no consistent knowledge on which type of peripheral sensory feedback may be effective in affecting the cortical plasticity or on how to best apply the sensory feedback.

The aim of the proposed research is to create natural, meaningful sensations through providing non-invasive sensory feedback (i.e. surface electrical stimulation) and the effectiveness to alleviate phantom limb pain and restore the cortical neuroplastic changes.

DETAILED DESCRIPTION:
Purpose of the experiment

Up to 50-80 % of persons with amputations experience pain in the part of the body that is missing. This phenomenon is called phantom limb pain. It is not clear today why phantom limb pain occurs, and since the pain can be difficult to treat, it can affect the quality of life. Other scientific studies have shown, that the use of electrical stimulation applied through surface electrodes, can assist to decrease or alleviate the phantom limb pain. The aim of this study is to investigate if daily surface electrical stimulation for a period of 30 days can decrease or alleviate the phantom limb pain.

Methods

Before the study begins, it will be necessary to test if the participant can tolerate the electrical stimulation and that the participant fulfill all criteria for participating in the study. During the study, different electrical stimulation sequences will be applied. The participant will be asked to fill out a series of questionnaires before, during and after the electrical stimulation, to describe how the electrical stimulation is experienced, and if the stimulation had an effect on the phantom limb pain and phantom sensations. The participant will also be asked about their general mood to investigate if this has an effect on the pain. The brain signals of the participants brain signals will be measured twice with either surface electrodes or with a scanning technique, while the participant is thinking about moving the amputated arm/hand or leg, while moving the healthy arm/leg, or while receiving electrical stimulation.

Plan for the experiment

The experiment will take place over a period of three months and consists of a series of measurement and intervention sessions planned in five phases. All sessions will take place at Aalborg University, Denmark except for the days when the brain signals are measured by using the scanning technique, which will take place at Aalborg University Hospital, Denmark.

Phase 1. Interview and meeting with the subject (before the experiment begins, 1 session, 1-2 hours). Before the experiment begins, the participant is invited to a meeting and interview with project responsible to inform the participant about the experiment.

Phase 2. Preliminary investigation (1 session of maximum 3 hours before the experiment starts). Before the experiment starts, but after the participant has signed the informed consent, the investigators will test if the participant can tolerate the electrical stimulation. If all criteria for participation are fulfilled, the participation of the subject will be decided.

Phase 3. Baseline measurements (day 1-27, 2 weekly sessions, maximum of 3 hours for each session). Before the repeated, electrical stimulation sessions begin, a series of baseline measurements will be performed. In this phase the sensory threshold (i.e., the level of the electrical stimulation that you can feel) will be measured, and the electrical stimulation parameters determined. The brain signals of the participant will be measured by a scanning technique (so-called functional magnetic resonance imaging or fMRI) and by surface electrodes placed oh the scalp (so-called electroencephalographic recordings or EEG). On the day that the brain signals are measured the session may last up to 5 hours.

Phase 4. Intervention period (day 28-56, 2-5 weekly sessions, maximum of 3 hours for each session). In these sessions, electrical stimulation will be applied through surface electrodes placed on the upper arm/the stump or the leg. The participant will be asked to fill out a series of questionnaires to report on the phantom limb pain, phantom sensations (i.e., non-painful sensations) and their general mood. Again the participant's brain signals will be measured using the scanning and the surface electrode techniques. On the day that the brain signals are measured the session may last up to 5 hours.

Phase 5. Follow-up (day 57-112, 4 weekly session over 8 weeks of maximum 3 hours). To measure the effect and duration of the intervention the participant will be asked to fill out a series of questionnaires.

Risks, side effects and disadvantages

Surface stimulation may cause muscle-contractions. Attachment of the surface electrodes may cause the skin to become red or irritated for some hours following the experiment. The type of electrical stimulation used in this experiment is not associated with any known risks or side effects. When the sensory threshold is determined (i.e., the lowest strength of the electrical stimulation that the participant can feel), it may feel unpleasant or painful for a short period of time, but the unpleasantness or pain will disappear as soon as the electrical stimulation stops. The electrical stimulation applied during the intervention period will be adjusted such that is it not painful.

Measurement of the brain signals using the fMRI-technique (scanning) is safe, and there are no known risks or side effects of this procedure. The participant may, however, find that being placed inside the scanner is unpleasant. Measurement of the brain signals with surface electrodes is also considered safe, and there are no known risks or side effects of this procedure. There may be risks associated with the experiment that are unknown to the investigators. Therefore, the participant is asked to inform the investigators if the participant experiences any health problems during the experiment. If the investigators discover any side effects, the participant will be informed immediately.

Benefits of the experiment

There will be no benefits for the subject by participation in the study. However, the participant may find that his/her phantom limb pain is alleviated during the experiment as a result of the electrical stimulation. However, it is not possible for the investigators to predict if the electrical stimulation will affect the phantom limb pain, when the effect will start, how large the effect will be, or how long the effect will last. It is not possible to offer the participants a permanent or lasting solution after termination of the study.

Exclusion from and suspension of the experiment

If the participant, according to the assessment of the investigator, react unexpectedly on the procedures or in any other way are not suitable for continuing in the experiment, the participation in the experiment can be terminated at any time. In general, the experiment will be terminated if it turns out that the subjects in general cannot tolerate the procedures of the project or find the experiment too exhausting.

ELIGIBILITY:
Inclusion Criteria:

* Amputation of one or both arms below the shoulder level or amputation of one or both legs below hip joint
* Total or partial peripheral nerve injury (i.e.,under spinal cord level) causing paralysis of the arms or legs
* Other treatments for phantom limb pain should have been tried with poor results
* The subject should experience phantom limb pain at a level of 6 or higher measured on on a visual analog scale (VAS) ranging from 0-10
* Phantom limb pain should be experienced at least once a week
* The subject should be in a chronic and stable phase, and the stump should have healed
* The subject should otherwise be healthy and able to carry out the experiment
* If pain medication is used it will be acceptable that the person continues to use the medication
* It should, through peripheral electrical stimulation, be possible to apply the relevant phantom emotions to the subject

Exclusion Criteria:

* Cognitive impairment
* Pregnancy
* Prior or current psychological diseases such as borderline, schizophrenia, depression or manic-depressive
* Acquired brain injury with residual impairment
* Prior neurological or musculoskeletal diseases
* History of or active substance abuse disorder
* Persons with that experience an allergic reaction to surface electrodes
* Persons with fear for electrical stimulation or pain
* Persons that are hypersensitive to electrical stimulation and experience the stimulation as unpleasant
* Persons that feel may claustrophobic in an MRI scanner
* Persons that have metal parts in the body (such as pacemakers or metal screws)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain | Change in pain perception over three months
  The pain intensity will be assessed using a visual analog scale (VAS)
Cortical reorganization | Change in cortical reorganization over three months
  The cortical response to peripheral stimulation will be tracked using MRI

SECONDARY OUTCOMES:
Cortical reorganization | Change in cortical reorganization over three months
  The cortical response to peripheral stimulation will be tracked using EEG
Phantom limb pain | Change in neuropathic pain symptoms over three months
  The pain symptoms wil be assessed using the neuropathic pain symptom inventory (NPSI)

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Jensen, Ph.D, Principal Investigator — Aalborg University
Locations (1):
- Winnie Jensen, Aalborg, Denmark